CLINICAL TRIAL: NCT04874805
Title: Oxygen Hemoglobin Saturation in COVID Patients: Comparison of Arterial Gasometry and Pulse Oximetry
Brief Title: Oxygen Saturation: Analytical Comparison for COVID
Acronym: SHOCOVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: since the departure of Dr. LEFRERE no investigator has decided to take over the project
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210142
Record Dates: First submitted 2021-04-16; First posted 2021-05-06 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hypoxemia; Covid-19
MeSH Terms: conditions — Hypoxia; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Major patient admitted to the ICU for COVID (Experimental)
  Interventions: Other: Measurement of oxygen saturation

INTERVENTIONS:
Other: Measurement of oxygen saturation — Measurement of oxygen saturation by pulse oximetry once a day, at 6 a.m., for a minimum of 3 days, thanks to three pulse oximeters (1 measurement point per device/day), in parallel with a synchronous sampling, programmed as part of the usual care, of arterial gasometry.

SUMMARY:
In many patients, respiratory Sars-Cov2 infection causes arterial hypoxemia, which remains without signs of verbalized respiratory distress, up to a point. This phenomenon, called "happy" or "silent" hypoxemia, has a plural pathophysiological basis. Hypoxemia has been shown to be predictively associated with admission to the ICU. Therefore, the question of constant monitoring of oxygenation, practiced on a large scale, at home, in asymptomatic patients or contact cases, arises. A large number of portable pulse oximeter are currently freely available on the market; however, their clinical validation remains sometimes doubtful, or even absent from FDA standards.

The objective of this study is to evaluate the accuracy of SpO2 values provided by portable pulse oximeter in COVID patients, in comparison with the reference method. The study will be conducted on a population of adult patients with COVID, hospitalized in the ICU, for whom gasometry sampling is already scheduled in the usual management.

DETAILED DESCRIPTION:
The constant monitoring of saturation by the pulse oximeter, the result of three centuries of technological progress, has introduced a true revolution in medical management that now relies on this vital parameter. In many patients, Sars-Cov2 respiratory infection causes arterial hypoxemia, which remains without signs of verbalized respiratory distress, up to a certain point. This phenomenon, called "happy" or "silent" hypoxemia, has a plural pathophysiological basis. Hypoxemia has been shown to be predictively associated with admission to the ICU. Therefore, the question of constant monitoring of oxygenation, practiced on a large scale, at home, in asymptomatic patients or contact cases, arises.

Despite its many advantages (non-invasive, kinetic), the pulse oximeter can be misused in several pathophysiological situations. The reference method for measuring hemoglobin oxygen saturation remains arterial gasometry.

However, a large number of portable pulse oximeter are currently freely available on the market; however, their clinical validation is sometimes questionable or even absent from FDA standards.

The objective of this study is to evaluate the accuracy of SpO2 values provided by portable pulse oximeter in COVID patients, in comparison with the reference method (arterial gasometry). The study will be conducted on a population of adult patients with COVID, hospitalized in the ICU, for whom gasometry sampling is already scheduled in the usual management.

Daily at 6am, during the systematic monitoring, arterial gasometry will be taken (as part of routine care) by the nurse or medical staff on duty. Synchronous measurement of Sp02 given by three portable pulse oximeter (1 measurement point per device, therefore 3 measurements/patient/day for a minimum of 3 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the intensive care unit for COVID
* Age ≥ 18 years
* Patients or family/trusted person informed and not objecting to participating in the research

Exclusion Criteria:

* Carbon monoxide poisoning
* Homozygous sickle cell disease
* Severe anemia (< 7 g/L) with associated hypoxemia
* Methemoglobinemia
* Sulfhemoglobinemia
* Sepsis, vasoconstrictive drugs
* Patients under guardianship / curators
* Patient under state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of SpO2 value provided by portable pulse oximeter in COVID patients compared with the reference method. | once a day
  Measurement of oxygen saturation by pulse oximetry once a day, at 6 a.m., for a minimum of 3 days, using three pulse oximeters (1 measurement point per device/day), in parallel with a synchronous, programmed arterial gasometry sampling Evaluation according to the standards of the SFBC (French Society of Clinical Biology) for the comparison of methods: minimum 40 points per apparatus, evenly distributed over the pathophysiological range of the saturations explored (9, 10): 60-100%.

SECONDARY OUTCOMES:
Identification of pathophysiological or analytical biases specific to COVID patients. | through study completion, an average of 7 months
  Data analysis will allow to identify potential biases in the measurement of oxygen saturation in COVID patients

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie, Médecine Intensive et Réanimation (SPMIR-R3S) Hôpital Pitié-Salpêtrière, Paris, France